CLINICAL TRIAL: NCT03871452
Title: Haydarpaşa Numune Education and Research Hospital
Brief Title: The Effectiveness of Ankaferd Blood Stopper in the Management of Traumatic Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, nazmiye koyuncu, specialist of emergency medicine, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: h8w67r3k
Record Dates: First submitted 2019-03-05; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Bleeding Disorder
Keywords: Ankaferd BloodStopper, laceration, bleeding
MeSH Terms: conditions — Hemostatic Disorders; Lacerations; Hemorrhage | interventions — ankaferd blood stopper

STUDY DESIGN:
Intervention Model Description: The study was conducted on patients with bleeding associated with extremity lacerations. All consecutive patients presented to the emergency department of the high-volume training hospital in Istanbul were recruited within the study period
Masking Description: I don't understand very well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABS in external bleeding (Active Comparator): Drug Ankaferd Blood Stopper Bleeding control in 10 minutes with ABS
  Interventions: Procedure: Ankaferd Blood Stopper in theTraumatic Bleeding
- Repetition of ABS stopped bleeding (Active Comparator): Repetition of ABS stopped bleeding
  Interventions: Procedure: Ankaferd Blood Stopper in theTraumatic Bleeding

INTERVENTIONS:
Procedure: Ankaferd Blood Stopper in theTraumatic Bleeding — ankaferd blood stpper They were trained to apply compression of approximately 3-kg weight after irrigation with saline in patients with active bleeding who met inclusion criteria. Bleeding was controlled in every minute and data were collected. Traditional methods such as primary suturing were performed in patients whose bleeding did not stop within 10 minutes. Patients whose bleeding was stopped were monitored for half an hour for bleeding recurrence.
  The patients were divided into two groups; ones treated by ABS soaked wet compresses (group I) and ones treated by dry sponge compresses

SUMMARY:
The objective of this study was to prospectively compare effectiveness of Ankaferd Blood Stopper (ABS) with dry sponges in cessation of bleeding in adult trauma cases with external bleeding due to extremity lacerations.

Methods: The study was conducted on patients with bleeding associated with extremity lacerations. All consecutive patients presented to the emergency department of the high-volume training hospital in Istanbul were recruited within the study period

DETAILED DESCRIPTION:
This study was planned as a prospective randomized study. After local ethics committee approval, all consecutive patients admitted to the Emergency Department of the Haydarpasa Numune Training & Research Hospital due to extremity lacerations between October 1st and October 11th 2018 were recruited. The longest duration for wound healing, infection follow-up, and suture removal was 12 days. Therefore, the study was completed in a total of 23 days after suture removal of the last case.

ABS which was approved in 2017 by the Ministry of Health, is being used routinely in the management of the patients with traumatic bleeding in the emergency department of the hospital. Nurses working in treatment areas of the department were trained for this prospective study. They were trained to apply compression of approximately 3-kg weight after irrigation with saline in patients with active bleeding who met inclusion criteria. Bleeding was controlled in every minute and data were collected. Traditional methods such as primary suturing were performed in patients whose bleeding did not stop within 10 minutes. Patients whose bleeding was stopped were monitored for half an hour for bleeding recurrence.

The patients were divided into two groups; ones treated by ABS soaked wet compresses (group I) and ones treated by dry sponge compresses (group II). Demographic data, systemic disease history, drugs used, injury mechanism, habits etc. of the patients enrolled in the study were recorded into data collection form.

Forty commercially prepared ABS-soaked wet sterile sponges and 40 dry sponges of 2.5x7 cm were randomly numbered and placed in a box in the study area. Random numbers table was used to generate the sequence of enumeration of the sponges. Any given patient was treated with the next sponge with the smallest number in the box and data sheets contained the number of the sponge with which the patient's bleeding was intervened. Therefore, allocation concealment was accomplished for the study purposes.

In both groups, lacerations that did not stop bleeding within 10 minutes and lacerations with recurred bleeding within the half-hour follow-up period were repaired by the primary suturing. Lacerations were sutured at the end of follow-up period in other patients. Daily dressing was recommended to the patients at discharge, and they were invited for a follow-up visit 3 days later. They were followed-up for wound infection. Suture removal date was recorded in data collection form.

Statistical analysis was conducted by using the MedCalc Statistical Software version 12.7.7 (MedCalc Software bvba, Ostend, Belgium; http://www.medcalc.org; 2013). Descriptive statistics were used to define continuous variables in this study (mean, standard deviation, range, and median). Mann Whitney U test was used to compare two independent and abnormally distributed groups. Chi-square test was performed to compare categorical variables, or Fisher's Exact test was performed where appropriate or required. Statistical significance level was determined as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years-old and above)
* presented with isolated cuts on the extremities
* cuts sized between 1 and 5 centimeters .

Exclusion Criteria:

* Patients under 18 years of age
* with only superficial abrasions
* with lacerations smaller than 1 cm and larger than 5 cm
* irregular laceration borders or star-like lacerations
* deep lacerations requiring subcutaneous suturing
* lacerations requiring additional interventions such as tendon repair controlled bleeding
* grade III and IV systemic diseases (advanced heart failure, uncontrolled hypertension, etc.) according to American Society of Anesthesiologists (ASA) classification,
* who received radiotherapy or chemotherapy for malignancies within the last three months
* with the history of hematologic diseases such as leukemia
* using medications leading to hemorrhage risk (oral anticoagulants, aspirin, etc.)
* congenital coagulation factor deficiency such as hemophilia
* multiple trauma and abnormal vital signs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Bleeding control | 1-10 minute
  Group I were compressed with ABS-soaked wet sponge, and group II were treated with compression using dry sterile sponges. The compresses were briefly removed at one-minute intervals and bleeding status were checked. This process was continued for a maximum of 10 minutes. The time when both stopped the bleeding was noted for comparison.The main issue here was to see how long the ABS had taken control of the bleeding
Repetition of bleeding | 0-30 minute
  Wounds were monitored for half an hour for bleeding recurrence

SECONDARY OUTCOMES:
Wound infection | 3-5 days
  They were invited for a follow-up visit 3 days later for wound infection

OTHER OUTCOMES:
Suture removal | 8-12 days
  Suture removal date was recorded in data collection form.

CONTACTS AND LOCATIONS:
Overall Officials: Cagatay Nuhoglu, MD, Principal Investigator — Haydarpasa Numune Education and Research Hospital/İSTANBUL/TURKEY
Locations (1):
- Nazmiye Koyuncu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beyazit Y, Kurt M, Kekilli M, Goker H, Haznedaroglu IC. Evaluation of hemostatic effects of Ankaferd as an alternative medicine. Altern Med Rev. 2010 Dec;15(4):329-36. PMID 21194248
- [Result] Goker H, Haznedaroglu IC, Ercetin S, Kirazli S, Akman U, Ozturk Y, Firat HC. Haemostatic actions of the folkloric medicinal plant extract Ankaferd Blood Stopper. J Int Med Res. 2008 Jan-Feb;36(1):163-70. doi: 10.1177/147323000803600121. PMID 18304416
- [Result] Ucar Albayrak C, Caliskan U, Haznedaroglu IC, Goker H. Haemostatic actions of the folkloric medicinal plant extract Ankaferd Blood Stopper. J Int Med Res 2008; 36:163-170. J Int Med Res. 2008 Nov-Dec;36(6):1447-8; author reply 1448-9. No abstract available. PMID 19094458
- [Result] Ozel Demiralp D, Haznedaroglu IC, Akar N. Functional proteomic analysis of Ankaferd(R) Blood Stopper. Turk J Haematol. 2010 Jun 5;27(2):70-7. doi: 10.5152/tjh.2010.03. PMID 27263447
- [Result] Tuncer I, Doganay L, Ozturk O. Instant control of fundal variceal bleeding with a folkloric medicinal plant extract: Ankaferd Blood Stopper. Gastrointest Endosc. 2010 Apr;71(4):873-5. doi: 10.1016/j.gie.2009.08.021. Epub 2009 Nov 17. No abstract available. PMID 19922917
- [Result] Ozaslan E, Purnak T, Yildiz A, Haznedaroglu IC. Bleeding due to slippage of elastic band during variceal ligation: successful use of Ankaferd blood stopper. Indian J Gastroenterol. 2010 Jul;29(4):166-8. doi: 10.1007/s12664-010-0043-y. Epub 2010 Sep 3. PMID 20814774
- [Result] Al B, Yildirim C, Cavdar M, Zengin S, Buyukaslan H, Kalender ME. Effectiveness of Ankaferd blood stopper in the topical control of active bleeding due to cutaneous-subcutaneous incisions. Saudi Med J. 2009 Dec;30(12):1520-5. PMID 19936413
- [Derived] Koyuncu N. The Effectiveness of Ankaferd Blood Stopper in the Management of Traumatic Bleeding. Adv Ther. 2019 May;36(5):1143-1149. doi: 10.1007/s12325-019-00935-4. Epub 2019 Mar 21. PMID 30900196